CLINICAL TRIAL: NCT03650322
Title: Effects of Yoga, Strength Training and Aerobic Exercise on Cognition in Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Neha P. Gothe, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18922
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Cancer; Cancer-related Problem/Condition; Exercise
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga Practice (Experimental): Participants will be led through a beginner yoga course taught by a certified yoga instructor. Classes will meet twice a week for 75 minutes each for the duration of 12 weeks. Sessions will focus on yoga postures, breathing, and meditative practices and may utilize mats, blocks, belts, and blankets.
  Interventions: Behavioral: Yoga
- Stretching and Toning (Active Comparator): This 12 week, progressive stretching and toning course will aid participants in building whole body strength and flexibility by utilizing weights, chairs, mats, and various other exercise equipment. Sessions will meet three times a week for 50 minutes and will offer 'easy' and 'hard' modifications taught by an exercise leader.
  Interventions: Behavioral: Stretching and Toning
- Aerobic Walking (Experimental): Participants will partake in treadmill walking that encourages them to reach a pre-determined heart rate range. Sessions will be conducted three times a week for 50 minutes, and offer participants to self-select a speed and incline to meet their target heart rate zone.
  Interventions: Behavioral: Aerobic Walking

INTERVENTIONS:
Behavioral: Yoga — 12 weeks, total of 150 minutes of exercise per week.
  Arms: Yoga Practice
Behavioral: Stretching and Toning — 12 weeks, total of 150 minutes of exercise per week.
  Arms: Stretching and Toning
Behavioral: Aerobic Walking — 12 weeks, total of 150 minutes of exercise per week.
  Arms: Aerobic Walking

SUMMARY:
The investigators propose to compare the effects of a 12-week, supervised, site-based group yoga intervention on cognitive function, functional fitness, and well-being in middle-aged cancer survivors. Subjects will be randomly assigned to one of three exercise conditions: a yoga group, an aerobic walking group or a strength training group. All sessions (2-3 times per week) will be led by a trained exercise leader for a total of 150 minutes of exercise each week for the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years of age
* Cancer diagnosis
* 1 year since last cancer treatment (surgery, chemotherapy, and/or radiation)
* Not planning to receive treatment during study period
* Completion of Physical Activity Readiness Questionnaire (PAR-Q)
* Ambulatory and absence of health conditions that may be exacerbated by yoga, walking, or strength training
* Physician consent (if deemed necessary)
* Low-active, i.e. less than 150 minutes/week of moderate to vigorous exercise, no current yoga practice (including within last six months)
* Intention to remain in the Champaign-Urbana area over the study duration
* Willingness to be randomly assigned to one of the three groups (yoga, aerobic walking, strength training)
* Comfortable with reading, writing, and speaking English

Exclusion Criteria:

* Below 30 or above 70 years of age
* Cancer diagnosis of the brain
* Less than 1 year since last treatment (surgery, chemotherapy, and/or radiation) or plans to receive treatment during study
* Determined ambulatory or 'high risk' based on responses to PAR-Q
* High-active (exercising more than 150 minutes/week in the last six months)
* No consent from physician
* Intent to be away from the Champaign-Urbana area for an extended period of time during the study
* Inability to communicate effectively in English

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Cognitive Function | Change from baseline to 12 weeks will be reported
  Participants will complete part of the NIH Toolbox measures that assess cognitive function.

SECONDARY OUTCOMES:
Cardiovascular Function | Change from baseline to 12 weeks will be reported
  Participants will complete a submaximal exercise test to reach a target heart rate within 85% of the age-predicted maximum.

OTHER OUTCOMES:
Feasibility: Recruitment and retention rates | Baseline to 12-weeks
  Proportion of participants randomized relative to total contacts, Proportion of participants who complete follow-up questionnaires,

CONTACTS AND LOCATIONS:
Overall Officials: Neha Gothe, Ph.D., M.A., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gothe NP, Erlenbach ED, Streeter SL, Lehovec L. Effects of yoga, aerobic, and stretching and toning exercises on cognition in adult cancer survivors: protocol of the STAY Fit pilot randomized controlled trial. Trials. 2020 Sep 15;21(1):792. doi: 10.1186/s13063-020-04723-2. PMID 32933561
- See also: Exercise Psychology Lab — http://epl.illinois.edu